CLINICAL TRIAL: NCT03313310
Title: Work-to-Prevent: Employment as HIV Prevention for Young Men Who Have Sex With Men (YMSM) and Young Transgender Women (YTW)
Brief Title: ATN 151 Work-to-Prevent: Employment as HIV Prevention
Acronym: W2P
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ATN 151; 5U24HD089880-02 (NIH)
Record Dates: First submitted 2017-09-20; First posted 2017-10-18 (Actual); Results first posted 2020-11-04 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: HIV Prevention
Keywords: Youth Empowerment; Employment Intervention; Young Men Who Have Sex With Men; Young Transgender Women

STUDY DESIGN:
Intervention Model Description: A single-arm longitudinal pre/post study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Employment Intervention (Experimental): An employment intervention (iFOUR) that has been adapted from previous piloting work of focus groups, key informant interviews and a community advisory board.
  Interventions: Behavioral: Employment Intervention

INTERVENTIONS:
Behavioral: Employment Intervention — Participants will complete 4 workshop sessions in groups of 6-12. The workshop curriculum was based on the pre-existing iFOUR program, and tailored based on feedback from a Community Advisory Board (CAB), Focus Groups, and In Depth Interviews.
  Other Names: iFOUR

SUMMARY:
The investigators aim to pilot-test a novel social and structural-level HIV intervention for YMSM and YTW of color ages 16-24.

DETAILED DESCRIPTION:
Work2Prevent will advance the science by adapting, tailoring, and pilot-testing a novel social and structural-level HIV intervention for YMSM and YTW of color ages16-24 aimed at increasing economic stability (i.e., employment) through youth empowerment and asset development, and decreasing HIV risk behaviors (i.e., sex work) associated with social and economic marginalization.

ELIGIBILITY:
Phase 2 Inclusion Criteria:

1. Being male or assigned male at birth (YTW)
2. Identifies as a man who has sex with men (YMSM) and/or a gay bisexual man or transgender woman/transwoman
3. Identifies as African American/Black or Hispanic/Latino
4. 16-24 years old
5. English-speaking (primary)
6. Currently unemployed but seeking employment, or employed only part-time (35 hrs or less on avg/wk)
7. Is able to attend a 4-session employment program

Phase 2 Exclusion Criteria:

1. Individuals identifying as non-Hispanic White
2. Individuals not assigned male at birth
3. Individuals with a known HIV positive-status at time of consent

Phase 3 Inclusion Criteria:

1. Being male or assigned male at birth (YTW)
2. Identifies as a man who has sex with men (YMSM) and/or a gay bisexual man or transgender woman/transwoman
3. Identifies as African American/Black or Hispanic/Latino
4. 16-24 years old
5. English-speaking (primary)
6. Currently unemployed but seeking employment, or employed only part-time (35 hrs or less on avg/wk)
7. Is able to attend a 4-session employment program
8. Did not participate in Phase 2

Phase 3 Exclusion Criteria:

1. Individuals identifying as non-Hispanic White
2. Individuals not assigned male at birth

Ages: 16 Years to 24 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Self-identifies as: (1) man who has sex with men (MSM) and/or gay or bisexual man or (2) transgender woman and/or transsexual male-to-female/transwoman.
Enrollment: 92 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2019-12-05 (Actual); Study Completion 2019-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brandon Hill, PhD, Principal Investigator — University of Chicago; Lisa Strader, MPH, Study Director — University of North Carolina, Chapel Hill
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified study data will be made available in the NICHD Data and Specimen Hub (DASH), a centralized resource for researchers to store de-identified data from NICHD supported studies for use in secondary research. NICHD DASH is a free public resource designed for the scientific research community.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be made available after data analyses have been completed, data has been de-identified, and all DASH submission requirements have been met and approved. Data will be available according to NICHD DASH timelines.
Access Criteria: Please see DASH guidelines for access criteria.
URL: https://dash.nichd.nih.gov/

REFERENCES:
- [Background] Barlow J., Wright C., Cullen L. A job-seeking self-efficacy scale for people with physical disabilities:preliminary development and psychometric testing. British Journal of Guidance and Counseling. 2002;30(1):37-53.
- [Background] Porter C., Woo S.E., Tak, J. Developing and Validating Short Form Protean and Boundaryless Career Attitudes Scales. Journal of Career Assessment. 2016;24(1):162-181.
- [Background] Horvath KJ, Oakes JM, Rosser BR, Danilenko G, Vezina H, Amico KR, Williams ML, Simoni J. Feasibility, acceptability and preliminary efficacy of an online peer-to-peer social support ART adherence intervention. AIDS Behav. 2013 Jul;17(6):2031-44. doi: 10.1007/s10461-013-0469-1. PMID 23553347
- [Background] Volmer J., Spurk D. Protean and boundaryless career attitudes: relationships with subjective and objective career success. 2011;43(3):207-218.
- [Derived] Hill BJ, Motley DN, Rosentel K, VandeVusse A, Fuller C, Bowers SME, Williams M, Kipke M, Kuhns L, Pashka N, Reisner S, DeMonte JB, Goolsby RW, Rupp BM, Slye N, Strader LC, Schneider JA, Razzano L, Garofalo R. Employment as HIV Prevention: An Employment Support Intervention for Adolescent Men Who Have Sex With Men and Adolescent Transgender Women of Color. J Acquir Immune Defic Syndr. 2022 Sep 1;91(1):31-38. doi: 10.1097/QAI.0000000000003020. Epub 2022 May 12. PMID 35551157
- [Derived] Hill BJ, Motley DN, Rosentel K, VandeVusse A, Garofalo R, Kuhns LM, Kipke MD, Reisner S, Rupp B, West Goolsby R, McCumber M, Renshaw L, Schneider JA. Work2Prevent, an Employment Intervention Program as HIV Prevention for Young Men Who Have Sex With Men and Transgender Youth of Color (Phase 3): Protocol for a Single-Arm Community-Based Trial to Assess Feasibility and Acceptability in a Real-World Setting. JMIR Res Protoc. 2020 Sep 11;9(9):e18051. doi: 10.2196/18051. PMID 32915162
- [Derived] Hill BJ, Motley DN, Rosentel K, VandeVusse A, Garofalo R, Schneider JA, Kuhns LM, Kipke MD, Reisner S, Rupp BM, Sanchez M, McCumber M, Renshaw L, Loop MS. An Employment Intervention Program (Work2Prevent) for Young Men Who Have Sex With Men and Transgender Youth of Color (Phase 1): Protocol for Determining Essential Intervention Components Using Qualitative Interviews and Focus Groups. JMIR Res Protoc. 2020 Aug 10;9(8):e16384. doi: 10.2196/16384. PMID 32773383
- [Derived] Hill BJ, Motley DN, Rosentel K, VandeVusse A, Garofalo R, Schneider JA, Kuhns LM, Kipke MD, Reisner S, Rupp BM, Sanchez M, McCumber M, Renshaw L, West Goolsby R, Loop MS. An Employment Intervention Program (Work2Prevent) for Young Men Who Have Sex With Men and Transgender Youth of Color (Phase 2): Protocol for a Single-Arm Mixed Methods Pilot Test to Assess Feasibility and Acceptability. JMIR Res Protoc. 2020 Aug 10;9(8):e16401. doi: 10.2196/16401. PMID 32773376

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants will be recruited in clinics serving young men who have sex with men (YMSM) and young transwomen (YTW) of color, and local gathering places for YMSM and YTW. Participants will be asked to refer potentially eligible friends or acquaintances. Passive recruitment will include posting study flyers and describing the study on social media.
Groups:
- Phase 2: Phase 2 utilizes a single-arm design, the intervention consists of four workshop sessions held over a two-week period.
- Phase 3: Phase 3 utilizes a single-arm design, the intervention consists of four workshop sessions held over a two-day period.
Period: Phase 2
Arm/Group | Phase 2 | Phase 3
Started | 51 | 0 (Phase 2 participants did not participate in Phase 3.)
Completed | 47 | 0 (Phase 2 participants did not participate in Phase 3.)
Not Completed | 4 | 0
Not completed — Lost to Follow-up | 4 | 0
Period: Phase 3
Arm/Group | Phase 2 | Phase 3
Started | 0 (Phase 3 participants did not participate in Phase 2.) | 41
Completed | 0 (Phase 3 participants did not participate in Phase 2.) | 40
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: The analysis population consists of participants who completed at least one workshop and/or the 8-month (3-month) follow-up visit.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 2 | Phase 3 | Total
Number analyzed (Participants) | 47 | 40 | 87
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 22 [19 to 23] | 22 [20 to 23.5] | 22 [20 to 23]
Sex/Gender, Customized [Count of Participants; unit: Participants] — self-identity; all individuals were assigned male sex at birth.
  Participants
    Female | 3 | 2 | 5
    Male | 35 | 23 | 58
    Transfemale or Transwoman | 6 | 11 | 17
    Transmale or Transman | 0 | 0 | 0
    Genderqueer or Gender Nonconforming | 3 | 4 | 7
    Other Gender Identity | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 4 | 15
  Not Hispanic or Latino | 36 | 36 | 72
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 41 | 38 | 79
  White | 1 | 0 | 1
  Other | 5 | 1 | 6
  American Indian or Alaskan Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants] — United States, Chicago
  Participants
    United States | 47 | 40 | 87
Sexual Orientation [Count of Participants; unit: Participants]
  Bisexual | 19 | 12 | 31
  Gay | 19 | 18 | 37
  Homosexual | 0 | 1 | 1
  Queer | 5 | 0 | 5
  Same Gender Loving | 0 | 2 | 2
  Straight or Heterosexual | 4 | 5 | 9
  Other | 0 | 2 | 2
Employment Status [Count of Participants; unit: Participants]
  Not Employed | 41 | 34 | 75
  Part-Time | 6 | 6 | 12
  Full-Time | 0 | 0 | 0
Job Seeking Self-Efficacy Score [Median (Inter-Quartile Range); unit: units on a scale] — Job seeking self-efficacy is defined as one's perceived ability and confidence to perform job search and application activities. The 12-item Job Seeking Self-Efficacy (JSS) scale uses response values on a 1-10 score, with 1 being "Not at All Confident" and 10 being "Very Confident". Responses are averaged to yield a total score, with higher scores indicating higher self-efficacy.
  units on a scale | 9.1 [7.9 to 10] | 8.5 [7.6 to 9.9] | 8.8 [7.8 to 10]
Baseline HIV Test Result [Count of Participants; unit: Participants] — Phase 3 participants who reported positive HIV status at baseline were not tested.
  Participants
    Reactive | 2 | 2 | 4
    Non-Reactive | 45 | 27 | 72
    Declined | 0 | 0 | 0
    HIV+ at Consent | NA — Known HIV positive status was an exclusion criterion for phase 2 only. | 11 | NA — Total not calculated because data are not available (NA) in one or more arms.
Self-Reported Sexual Risk Behaviors [Number; unit: Number of events] — Note that Self-Reported Sexual Risk Behaviors are not mutually exclusive categories.
  Abbreviations: CAI, Condomless anal intercourse; STI, sexually transmitted infection.
  Number of events
    CAI with Male Partner of Unknown HIV Status | 12 | 9 | 21
    Anal Intercourse with 3 or More Male Partners | 23 | 21 | 44
    Sex with Male Partner with STI | 6 | 11 | 17
    CAI with HIV+ Male Partner | 8 | 10 | 18
    Anal Intercourse with Condom Failure | 10 | 14 | 24
    Transactional Sex Work Involvement | 15 | 21 | 36
Number of Self-Reported Sexual Risk Behaviors [Count of Participants; unit: Participants]
  0 Criteria | 16 | 8 | 24
  1 Criterion | 9 | 8 | 17
  2 Criteria | 11 | 8 | 19
  3 Criteria | 5 | 7 | 12
  4+ Criteria | 6 | 9 | 15

OUTCOME MEASURES:

1. Primary Outcome: Information Systems Success Model Score
Description: The Information Systems Success Model (ISSM) will be used to assess for intervention acceptability and satisfaction. The 21-item scale measures four sub-domains: information quality, handbook quality, perceived usefulness, and overall satisfaction. Every item is scored on a 1-5 scale, with 1 being "Strongly Disagree" and 5 being "Strongly Agree". Responses are averaged within each sub-domain to produce four sub-domain scores. The four sub-domain scores are then averaged to produce an overall ISSM score (1-5; higher scores indicate higher acceptability/satisfaction).
Time Frame: Post-Intervention (up to 2 weeks after completion of intervention)
Population: The analysis population consists of all participants who completed the post-intervention evaluation.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Phase 2 | Phase 3
Number analyzed (Participants) | 33 | 37
units on a scale | 4.4 [4.0 to 4.8] | 4.2 [3.8 to 4.7]

2. Primary Outcome: Number of Participants Completing Two or More Workshop Sessions
Description: Workshop completion will be used to assess for intervention feasibility, as the workshop sessions are the intervention. Workshop completion will be defined as having attended at least two of the four workshop sessions and will be measured by tracking participant attendance.
Time Frame: Post-Intervention (up to 2 weeks after completion of intervention)
Population: The analysis population consists of participants who completed at least one workshop and/or the 8-month follow-up visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2 | Phase 3
Number analyzed (Participants) | 47 | 40
Participants | 28 | 34

3. Primary Outcome: Change From Baseline in Job Seeking Self-Efficacy Scale Score
Description: Job seeking self-efficacy is defined as one's perceived ability and confidence to perform job search and application activities. The 12-item Job Seeking Self-Efficacy (JSS) scale uses response values on a 1-10 score, with 1 being "Not at All Confident" and 10 being "Very Confident". Responses are averaged to yield a total score, with higher scores indicating higher self-efficacy. Change in JSS will be calculated by subtracting the JSS score at baseline (T1) from the JSS score at the 8-month follow-up (T3) (-9 to +9; negative change indicates decreased self-efficacy, while positive change indicates increased self-efficacy).
Time Frame: Baseline, Follow-Up (8 months for Phase 2, 3 months for Phase 3)
Population: The phase 2 (phase 3) analysis population consists of participants who completed at least one workshop and/or the 8-month (3-month) follow-up visit. Participants with missing data at baseline and/or follow-up were excluded from the analysis.
Measure: Mean (90% Confidence Interval); unit: units on a scale
Arm/Group | Phase 2 | Phase 3
Number analyzed (Participants) | 46 | 40
units on a scale | -0.08 [-0.41 to 0.26] | 0.62 [0.14 to 1.11]
Statistical Analysis 1: Comparison: Phase 2; Test type: Other — A one-sample non-parametric test for change between baseline and 8-month follow-up was conducted; p = 0.98, Wilcoxon Signed Rank — The a priori threshold for statistical significance was set at 0.10. This p-value was not adjusted for multiple comparisons
Statistical Analysis 2: Comparison: Phase 3; Test type: Other — A one-sample non-parametric test for change between baseline and 3-month follow-up was conducted; p = 0.05, Wilcoxon Signed Rank — [p-value comment as in outcome 3, analysis 1]

4. Primary Outcome: Change From Baseline in Protean Career Attitudes Scale Score
Description: Protean career attitudes (PCAs) are defined as having self-direction in the pursuit of success in one's work. PCAs have previously been found to be associated with positive career satisfaction and self-perceived success. The validated 7-item scale measures two sub-domains: self-directed attitudes and values-driven attitudes. Every item is scored on a 1-5 scale, with 1 being "Strongly Disagree" and 5 being "Strongly Agree". Responses are averaged within each sub-domain to produce two sub-domain scores, which are then averaged as well to produce an overall PCA score. Change in PCA score will be calculated by subtracting the score at baseline (T1) from the score at the 8-month follow-up (T3) (-4 to +4; negative change indicates decreased PCAs, while positive change indicates increased PCAs).
Time Frame: Baseline, Follow-Up (8 months for Phase 2, 3 months for Phase 3)
Population: as for outcome 3
Measure: Mean (90% Confidence Interval); unit: units on a scale
Arm/Group | Phase 2 | Phase 3
Number analyzed (Participants) | 44 | 38
units on a scale | -0.09 [-0.25 to 0.06] | -0.03 [-0.27 to 0.21]
Statistical Analysis 1: Comparison: Phase 2; Test type: Other — A one-sample non-parametric test for change between baseline and 8-month follow-up was conducted; p = 0.39, Wilcoxon Signed Rank — [p-value comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Phase 3; Test type: Other — A one-sample non-parametric test for change between baseline and 3-month follow-up was conducted; p = 0.76, Wilcoxon Signed Rank — [p-value comment as in outcome 3, analysis 1]

5. Secondary Outcome: Change From Baseline in Self-Reported Hours Worked Per Week
Description: Employment status will be assessed using self-reported average number of hours worked each week. Change in hours worked per week will be calculated by subtracting the baseline (T1) value from the follow-up (T3) value (negative change indicates fewer hours worked per week, while positive change indicates more hours work per week).
Time Frame: Baseline, Follow-Up (8 months for Phase 2, 3 months for Phase 3)
Population: as for outcome 3
Measure: Mean (90% Confidence Interval); unit: hours/week
Arm/Group | Phase 2 | Phase 3
Number analyzed (Participants) | 43 | 37
hours/week | 11.4 [7.14 to 15.65] | 5.24 [1.54 to 8.94]
Statistical Analysis 1: Comparison: Phase 2; Test type: Other — A one-sample non-parametric test for change between baseline and 8-month follow-up was conducted; p < 0.001, Wilcoxon Signed Rank — [p-value comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Phase 3; Test type: Other — A one-sample non-parametric test for change between baseline and 3-month follow-up was conducted; p = 0.02, Wilcoxon Signed Rank — [p-value comment as in outcome 3, analysis 1]

6. Secondary Outcome: Change From Baseline in Self-Reported Sexual Risk Behaviors
Description: Sexual risk behaviors will be measured using 6 yes/no items assessing for engagement in the following behaviors during the past 6 months (this refers to the 6 months prior to the baseline visit for the first assessment and 6 months prior to the 8 month visit for the second assessment) for Phase 2, and the last 3 months for Phase 3:
  1. condomless anal intercourse (CAI) with male partner of unknown HIV status
  2. anal intercourse with 3 or more males
  3. sex with male partner with a Sexually Transmitted Infection (STI)
  4. CAI with HIV+ male partner
  5. anal intercourse with condom failure
  6. transactional sex work involvement
  Responses will be averaged at each assessment. Change in sexual risk behaviors will be calculated by subtracting the average at baseline from the average at the 8-month follow-up (range: -1 to +1; negative change indicates fewer sexual risk behaviors, while positive change indicates more sexual risk behaviors).
Time Frame: Baseline, Follow-Up (8 months for Phase 2, 3 months for Phase 3)
Population: as for outcome 3
Measure: Mean (90% Confidence Interval); unit: sexual risk factors
Arm/Group | Phase 2 | Phase 3
Number analyzed (Participants) | 44 | 38
sexual risk factors | -0.03 [-0.10 to 0.05] | -0.06 [-0.13 to 0.01]
Statistical Analysis 1: Comparison: Phase 2; Test type: Other — A one-sample non-parametric test for change between baseline and 8-month follow-up was conducted; p = 0.51, Wilcoxon Signed Rank — [p-value comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Phase 3; Test type: Other — A one-sample non-parametric test for change between baseline and 3-month follow-up was conducted; p = 0.17, Wilcoxon Signed Rank — [p-value comment as in outcome 3, analysis 1]

7. Secondary Outcome: Change From Baseline in Oral Chlamydia Test Result
Description: Chlamydia infection will be assessed at baseline and follow-up using an oral sample. The test yields a positive (1) or negative (0) result. The number of positive test results at baseline and follow-up will be calculated.
Time Frame: Baseline, Follow-Up (8 months for Phase 2, 3 months for Phase 3)
Population: The phase 2 (phase 3) analysis population consists of participants who completed at least one workshop and/or the 8-month (3-month) follow-up visit. 2 phase 2 participants who declined testing were excluded. 10 phase 2 and 8 phase 3 participants whose test results were missing, not collected, or unknown at baseline and/or follow-up were excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2 | Phase 3
Number analyzed (Participants) | 35 | 32
Participants
  Number of Positive Test Results at Baseline | 2 | 1
  Number of Positive Test Results at Follow-up | 0 | 0
Statistical Analysis 1: Comparison: Phase 2; Test type: Other; A one-sample McNemar's test for change between baseline and 8-month follow-up was planned. The a priori threshold for statistical significance was set at 0.10. However, McNemar's test statistic could not be calculated due to small cell counts
Statistical Analysis 2: Comparison: Phase 3; Test type: Other; A one-sample McNemar's test for change between baseline and 3-month follow-up was planned. The a priori threshold for statistical significance was set at 0.10. However, McNemar's test statistic could not be calculated due to small cell counts

8. Secondary Outcome: Change From Baseline in Anal Chlamydia Test Result
Description: Chlamydia infection will be assessed at baseline and follow up using an anal sample. The test yields a positive (1) or negative (0) result. Number of positive test results at baseline and follow-up will be calculated.
Time Frame: Baseline, Follow-Up (8 months for Phase 2, 3 months for Phase 3)
Population: The phase 2 (phase 3) analysis population consists of those who completed at least one workshop and/or the 8-month (3-month) follow-up. 1 phase 2 and 1 phase 3 participant who declined testing were excluded. 18 phase 2 and 8 phase 3 participants whose test results were missing, not collected, or unknown at baseline and/or follow-up were excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2 | Phase 3
Number analyzed (Participants) | 28 | 31
Participants
  Number of Positive Test Results at Baseline | 2 | 0
  Number of Positive Test Results at Follow-up | 3 | 2
Statistical Analysis 1: Comparison: Phase 2; Test type: Other — A one-sample test for change between baseline and 8-month follow-up was conducted; p = 1.00, McNemar — [p-value comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Phase 3; Test type: Other — A one-sample test for change between baseline and 3-month follow-up was conducted; p = 0.50, McNemar — [p-value comment as in outcome 3, analysis 1]

9. Secondary Outcome: Change From Baseline in Urine Chlamydia Test Result
Description: Chlamydia infection will be assessed at baseline and follow up using a urine sample. The test yields a positive (1) or negative (0) result. Number of positive test results at baseline and follow-up will be calculated.
Time Frame: Baseline, Follow-Up (8 months for Phase 2, 3 months for Phase 3)
Population: The phase 2 (phase 3) analysis population consists of participants who completed at least one workshop and/or the 8-month (3-month) follow-up visit. 1 phase 2 participant who declined testing was excluded. 12 phase 2 and 5 phase 3 participants whose test results were missing, not collected, or unknown at baseline and/or follow-up were excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2 | Phase 3
Number analyzed (Participants) | 34 | 35
Participants
  Number of Positive Test Results at Baseline | 1 | 2
  Number of Positive Test Results at Follow-up | 3 | 1
Statistical Analysis 1: Comparison: Phase 2; Test type: Other — A one-sample test for change between baseline and 8-month follow-up was conducted; p = 0.63, McNemar — [p-value comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Phase 3; Test type: Other — A one-sample test for change between baseline and 3-month follow-up was conducted; p = 1.00, McNemar — [p-value comment as in outcome 3, analysis 1]

10. Secondary Outcome: Change From Baseline in Oral Gonorrhea Test Result
Description: Gonorrhea infection will be assessed at baseline and follow-up using an oral sample. The test yields a positive (1) or negative (0) result. Number of positive test results at baseline and follow-up will be calculated.
Time Frame: Baseline, Follow-Up (8 months for Phase 2, 3 months for Phase 3)
Population: The phase 2 (phase 3) analysis population consists of participants who completed at least one workshop and/or the 8-month (3-month) follow-up. 2 phase 2 participants who declined testing were excluded. 10 phase 2 and 9 phase 3 participants whose test results were missing, not collected, or unknown at baseline and/or follow-up were excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2 | Phase 3
Number analyzed (Participants) | 35 | 31
Participants
  Number of Positive Test Results at Baseline | 2 | 3
  Number of Positive Test Results at Follow-up | 1 | 0
Statistical Analysis 1: Comparison: Phase 2; Test type: Other — A one-sample test for change between baseline and 8-month follow-up was conducted; p = 1.00, McNemar — [p-value comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Phase 3; Test type: Other — A one-sample test for change between baseline and 3-month follow-up was conducted; p = 0.25, McNemar — [p-value comment as in outcome 3, analysis 1]

11. Secondary Outcome: Change From Baseline in Anal Gonorrhea Test Result
Description: Gonorrhea infection will be assessed at baseline and follow-up using an anal sample. The test yields a positive (1) or negative (0) result. Number of positive test results at baseline and follow-up will be calculated.
Time Frame: Baseline, Follow-Up (8 months for Phase 2, 3 months for Phase 3)
Population: The phase 2 (phase 3) analysis population consists of those who completed at least one workshop and/or the 8-month (3-month) follow-up. 1 phase 2 and 2 phase 3 participants who declined testing were excluded. 17 phase 2 and 7 phase 3 participants whose test results were missing, not collected, or unknown at baseline and/or follow-up were excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2 | Phase 3
Number analyzed (Participants) | 29 | 31
Participants
  Number of Positive Test Results at Baseline | 3 | 2
  Number of Positive Test Results at Follow-up | 2 | 1
Statistical Analysis 1: Comparison: Phase 2; Test type: Other — A one-sample test for change between baseline and 8-month follow-up was conducted; p = 1.00, McNemar — [p-value comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Phase 3; Test type: Other — A one-sample test for change between baseline and 3-month follow-up was conducted; p = 1.00, McNemar — [p-value comment as in outcome 3, analysis 1]

12. Secondary Outcome: Change From Baseline in Urine Gonorrhea Test Result
Description: as for outcome 10
Time Frame: Baseline, Follow-Up (8 months for Phase 2, 3 months for Phase 3)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2 | Phase 3
Number analyzed (Participants) | 34 | 35
Participants
  Number of Positive Test Results at Baseline | 1 | 0
  Number of Positive Test Results at Follow-up | 0 | 0
Statistical Analysis 1: Comparison: Phase 2; Test type: Other; [other analysis details as in outcome 7, analysis 1]
Statistical Analysis 2: Comparison: Phase 3; Test type: Other; [other analysis details as in outcome 7, analysis 2]

13. Secondary Outcome: Reactive HIV Result or Reported New HIV+ Status
Description: HIV infection will be assessed at follow-up using reactive HIV testing. Test results yield: Reactive or Non-reactive. Participants who reported HIV+ status will not be tested. A reactive HIV result will be defined as those with a "Reactive" result. Reported new HIV+ status is defined as those who report positive HIV status at follow-up and who were tested for HIV, with a non-reactive result, at baseline.
Time Frame: Follow-Up (8 months for Phase 2, 3 months for Phase 3)
Population: The phase 2 (phase 3) analysis population consists of those who completed at least one workshop and/or the 8-month (3-month) follow-up. Participants with missing data at either time point were excluded from the analysis. Participants who reported HIV+ status were not tested.
  Two phase 3 participants reported new HIV+ status at follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2 | Phase 3
Number analyzed (Participants) | 37 | 24
Participants | 0 | 2

14. Post Hoc Outcome: Change From Baseline in Any Self-reported Condomless Anal Intercourse
Description: Self-reported condomless anal intercourse will be measured using 2 yes/no items assessing for engagement in the following behaviors during the past 6 months (this refers to the 6 months prior to the baseline visit for the first assessment and 6 months prior to the 8 month visit for the second assessment) for Phase 2, and the last 3 months for Phase 3:
  1. CAI with male partner of unknown HIV status
  2. CAI with HIV+ male partner
  Number of yes responses at baseline and follow-up will be calculated.
Time Frame: Baseline, Follow-Up (8 months for Phase 2, 3 months for Phase 3)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2 | Phase 3
Number analyzed (Participants) | 44 | 38
Participants
  Number of Yes Responses at Baseline | 14 | 13
  Number of Yes Responses at Follow-up | 13 | 12
Statistical Analysis 1: Comparison: Phase 2; Test type: Other — A one-sample test for change between baseline and 8-month follow-up was conducted; p = 1.00, McNemar — [p-value comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Phase 3; Test type: Other — A one-sample test for change between baseline and 3-month follow-up was conducted; p = 1.00, McNemar — [p-value comment as in outcome 3, analysis 1]

15. Post Hoc Outcome: Change From Baseline in Self-reported Sex With Male Partner With a Sexually Transmitted Infection
Description: Self-reported sex with a male partner with a sexually transmitted infection during the past 6 months (this refers to the 6 months prior to the baseline visit for the first assessment and 6 months prior to the 8 month visit for the second assessment) for Phase 2, and the last 3 months for Phase 3, will be measured using a yes/no item. Number of yes responses at baseline and follow-up will be calculated.
Time Frame: Baseline, Follow-Up (8 months for Phase 2, 3 months for Phase 3)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2 | Phase 3
Number analyzed (Participants) | 44 | 37
Participants
  Number of Yes Responses at Baseline | 5 | 11
  Number of Yes Responses at Follow-up | 5 | 9
Statistical Analysis 1: Comparison: Phase 2; Test type: Other — A one-sample test for change between baseline and 8-month follow-up was conducted; p = 1.00, McNemar — [p-value comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Phase 3; Test type: Other — A one-sample test for change between baseline and 3-month follow-up was conducted; p = 0.75, McNemar — [p-value comment as in outcome 3, analysis 1]

16. Post Hoc Outcome: Change From Baseline in Self-reported Anal Intercourse With Condom Failure
Description: Self-reported anal intercourse where the condom broke or slipped during the past 6 months (this refers to the 6 months prior to the baseline visit for the first assessment and 6 months prior to the 8 month visit for the second assessment) for Phase 2, and the last 3 months for Phase 3, will be measured using a yes/no item. Number of yes responses at baseline and follow-up will be calculated.
Time Frame: Baseline, Follow-Up (8 months for Phase 2, 3 months for Phase 3)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2 | Phase 3
Number analyzed (Participants) | 44 | 38
Participants
  Number of Yes Responses at Baseline | 9 | 14
  Number of Yes Responses at Follow-up | 12 | 15
Statistical Analysis 1: Comparison: Phase 2; Test type: Other — A one-sample test for change between baseline and 8-month follow-up was conducted; p = 0.55, McNemar — [p-value comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Phase 3; Test type: Other — A one-sample test for change between baseline and 3-month follow-up was conducted; p = 1.00, McNemar — [p-value comment as in outcome 3, analysis 1]

17. Post Hoc Outcome: Change From Baseline in Self-reported Transactional Sex Work Involvement
Description: Self-reported transactional sex work involvement during the past 6 months (this refers to the 6 months prior to the baseline visit for the first assessment and 6 months prior to the 8 month visit for the second assessment) for Phase 2, and the last 3 months for Phase 3, will be measured using a yes/no item. Number of yes responses at baseline and follow-up will be calculated.
Time Frame: Baseline, Follow-Up (8 months for Phase 2, 3 months for Phase 3)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2 | Phase 3
Number analyzed (Participants) | 44 | 38
Participants
  Number of Yes Responses at Baseline | 13 | 21
  Number of Yes Responses at Follow-up | 10 | 15
Statistical Analysis 1: Comparison: Phase 2; Test type: Other — A one-sample test for change between baseline and 8-month follow-up was conducted; p = 0.45, McNemar — [p-value comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Phase 3; Test type: Other — A one-sample test for change between baseline and 3-month follow-up was conducted; p = 0.07, McNemar — [p-value comment as in outcome 3, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the baseline through study completion, approximately 8 months for Phase 2 and 3 months for Phase 3.
Description: In addition to adverse events, untoward event data were collected, and are defined as unexpected occurrences involving study participants, study staff, or the community where the study is taking place, that may reasonably be judged as related to study procedures and that lead to harm, distress, or increased risk of harm or distress, but that do not otherwise meet the definition of an adverse event.
Arm/Group | Phase 2 | Phase 3
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/41
Other Adverse Events (participants affected / at risk) | 0/51 | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-08-05): https://cdn.clinicaltrials.gov/large-docs/10/NCT03313310/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-13): https://cdn.clinicaltrials.gov/large-docs/10/NCT03313310/SAP_001.pdf